CLINICAL TRIAL: NCT06195449
Title: Clinical and Radiographic Evaluation of Alkasite Restorative Material Versus Glass Ionomer Cement in Restoration of Primary Molars: Randomized Clinical Trial.
Brief Title: Clinical and Radiographic Evaluation of Alkasite Restorative Material Versus Glass Ionomer Cement
Acronym: GIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ola Yasir Abdulaziz Mahmoud, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: alkasite material
Record Dates: First submitted 2023-12-23; First posted 2024-01-08 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Tooth Decay
Keywords: Alkasite restorative material; cention N; GIC; Primary molars
MeSH Terms: conditions — Dental Caries | interventions — Glass Ionomer Cements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alkasite restorative material in primary molar (Experimental): ARM 1 : ALKASITE RESTORATIVE MATERIAL( INTERVENTION)
  Interventions: Other: ALKASITE RESTORATIVE MATERIAL
- Glass Ionomer Cement in primary molar (Active Comparator): ARM2: Glass Ionomer Cement(CONTROL)
  Interventions: Other: Glass Ionomer Cement

INTERVENTIONS:
Other: ALKASITE RESTORATIVE MATERIAL — Restorative material for primary teeth
  Other Names: cention n
  Arms: Alkasite restorative material in primary molar
Other: Glass Ionomer Cement — Restorative material for primary teeth
  Other Names: GIC
  Arms: Glass Ionomer Cement in primary molar

SUMMARY:
To evaluate the clinical and radiographic performance of Alkasite restorative material versus glass ionomer in restoration of primary molars.

DETAILED DESCRIPTION:
Restorations replacements are mostly caused by the existence of caries lesions surrounding the restorations, which are commonly referred to as secondary caries .

Secondary or recurrent caries is characterized as "lesions that occur at the edges of previously placed dental restorations" or "caries that develop in association with dental restorations or sealants" (CARS).Proper seal at the tooth surface restoration interface is essential . That's why the most frequently material used is (GIC) with the advantage of chemical adhesion to tooth structure, superior esthetics, and long-term fluoride release providing cariostatic effect, but it has the disadvantage of slow setting rate, low fracture toughness, susceptibility to moisture contamination, dehydration during initial phase of setting, and poor wear resistance.

Resin Modified Glass Ionomer and Composite have always been the preferred material for restoration although several modifications have been made recently to improve its properties, Cent ion N is one of the recent ones.

Cent ion N is a tooth-colored basic filling material for direct restoration. It belongs to the material of Alka sites, with high flexural strength. It also has calcium and fluoride releasing properties comparable to conventional GIC, besides it is quick and easy to use.

ELIGIBILITY:
Inclusion Criteria:

* 1. Children having carious primary molars without pulp exposure and normal radiograph.

  2. Children between age 5 and 7 years. 3. Both male and female are included. 4. Cooperative Children.

Exclusion Criteria:

* 1. Patients with systemic diseases. 2. Parent refuse to participate.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
recurrent caries of the tooth | 12 months
  Radiograph &Visual inspection using Modified United States Public Health Service Ryge criteria (USPHS

SECONDARY OUTCOMES:
Color match of the restoration | 12 months
  Visual Inspection using Modified United States Public Health Service Ryge criteria (USPHS)
Marginal Discoloration of the tooth | 12 months
  by Visual Inspection using Modified United States Public Health Service Ryge criteria (USPHS)
Marginal Adaptation of the tooth | 12 months
  by Visual Inspection and Explorer using Modified United States Public Health Service Ryge criteria (USPHS)
Anatomic Form of the tooth | 12 months
  by Visual Inspection and Explorer using Modified United States Public Health Service Ryge criteria (USPHS)

CONTACTS AND LOCATIONS:
Overall Officials: Sherien Ezz Eldin, Professor, Study Director — cairo university faculty of pediatric dentistry

IPD SHARING:
Plan to Share IPD: Yes
study protocol and statistical analysis
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after one year
Access Criteria: with other investigator including who will work with systematic review , will provide the clinical study report with the documents above

REFERENCES:
- [Background] Sharma H, Suprabha BS, Shenoy R, Rao A, Kotian H. Clinical effectiveness of alkasite versus nanofilled resin composite in the restoration of occlusal carious lesions in permanent molar teeth of children: a randomized clinical trial. Eur Arch Paediatr Dent. 2023 Jun;24(3):301-311. doi: 10.1007/s40368-023-00788-0. Epub 2023 Mar 22. PMID 36947344
- [Background] Hegazi, R.I., W.E. Jamil, and A. Fawzy, Comparative Evaluation of Clinical Performance of Three Different Glass Hybrid Restorations in High Caries Risk Patients: A Randomized Control Trial. Dental Science Updates, 2023. 4(1): p. 171-183.
- [Background] Bepu, D., et al., Alksite-based material to restore endodontically treated teeth: A randomized controlled clinical trial. 2023.
- [Background] Pooja MP, Karuna YM, Rao A, Suman E, Natarajan S, Suprabha BS. Comparative Evaluation of the Sealing Ability of an Alkasite Restorative Material and Resin-Modified Glass Ionomer Cement in Primary Molars: An In vivo Study. Contemp Clin Dent. 2022 Apr-Jun;13(2):113-117. doi: 10.4103/ccd.ccd_345_20. Epub 2022 Jun 21. PMID 35846588
- [Background] 9. Derchi, G., et al., Clinical Performance of CentionTM Alkasite Restorative Material vs. Glass Ionomer Cement Used in Deciduous Teeth: One-Year Evaluation. Applied Sciences, 2022. 12(21): p. 10845.
- [Background] 8. Attia, R., et al., Clinical Performance of Alkasite Dental Material and High Viscosity Glass Ionomer Restorations in Class I Cavities. Comparative Study for One Year Follow Up. Egyptian Dental Journal, 2022. 68(4): p. 3881-3894.
- [Background] Arora D, Jain M, Suma Sogi HP, Shahi P, Gupta I, Sandhu M. In vivo evaluation of clinical performance of Cention N and glass ionomer cement in proximal restorations of primary molars. J Indian Soc Pedod Prev Dent. 2022 Jan-Mar;40(1):23-29. doi: 10.4103/jisppd.jisppd_108_21. PMID 35439879
- [Background] Mushtaq U, Mushtaq F, Thakur D, Rathee K, Poonia N, Khullar S. Comparative Evaluation of Postoperative Sensitivity Following Restoration of Class I Lesions with Different Restorative Materials: An In Vivo Study. J Contemp Dent Pract. 2021 Jun 1;22(6):650-654. PMID 34393122
- [Background] 5. Minocha, A., et al., Comparative evaluation of Cention N and Amalgam in Class II posterior restorations. UNIVERSITY JOURNAL OF DENTAL SCIENCES, 2021. 7(1).
- [Background] 4. Roulet, J., et al., In vitro wear of two bioactive composites and a glass ionomer cement. DZZ International, 2019. 1(1): p. 24-30.
- [Background] 3. Dodiya, P.V., et al., Clinical evaluation of cention-n and nano hybrid composite resin as a restoration of noncarious cervical lesion. J Dent Specialities, 2019. 7(1): p. 3-5.
- [Background] 2. Modified United States Public Health Service (USPHS) Ryge Criteria for Direct Clinical Evaluation of Restoration. 1995.
- [Background] 1. Class, V., Comparative evaluation of microleakage of three different restorative materials (Cention N, Zirconomer improved and Glass hybrid restorative system) in Class V cavity restoration using stereomicroscope: In vitro study.